CLINICAL TRIAL: NCT01944007
Title: Open-label Phase 1 Multiple Dose Escalation Trial to Assess the Safety, Tolerability, and Efficacy of Capsules Containing Cross-linked Polyelectrolyte (CLP) Given to Normal Healthy Volunteers
Brief Title: Evaluation of Cross-Linked Polyelectrolyte (CLP) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sorbent Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CTST-5
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Basic Science: Safety, Tolerability, Efficacy of CLP
Keywords: CLP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CLP 15 g Fed (Experimental): Cross-Linked Polyelectrolyte (CLP) Study medication delivered q.i.d just before each of 4 standardized meals/snack
  Interventions: Drug: Cross-Linked Polyelectrolyte (CLP)
- CLP 25 g Fed (Experimental): Cross-Linked Polyelectrolyte (CLP) Study medication delivered q.i.d just before each of 4 standardized meals/snack
  Interventions: Drug: Cross-Linked Polyelectrolyte (CLP)
- CLP 7.5 g Fed (Experimental): Cross-Linked Polyelectrolyte (CLP) Study medication delivered q.i.d just before each of 4 standardized meals/snack
  Interventions: Drug: Cross-Linked Polyelectrolyte (CLP)
- CLP 15 g fasted (Experimental): Cross-Linked Polyelectrolyte (CLP) Study medication delivered q.i.d 1 hour prior to 4 standardized meals/snack
  Interventions: Drug: Cross-Linked Polyelectrolyte (CLP)

INTERVENTIONS:
Drug: Cross-Linked Polyelectrolyte (CLP) — CLP was administered orally, in capsules, for 9 consecutive days.

SUMMARY:
This is a dose-escalation study to determine the effect of CLP in normal healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females between the ages of 18 and 70 years
* Body mass index (BMI) between 18 and 32 kg/m^2, inclusive
* Females could not be pregnant or breast feeding and had to be using birth control

Exclusion Criteria:

* Positive drug screen for substances of abuse
* Positive results for HIV, hepatitis B, or hepatitis C
* Screening 12-lead ECG demonstrating QTc interval >430 msec for males and >450 msec for females, or any cardiac rhythm disorder considered by the Investigator to be clinically relevant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-12; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Net Sodium Balance | Days 5 - 9
  Daily net sodium balance was calculated based on dietary and fluid intake, urinary and fecal output and emesis.

SECONDARY OUTCOMES:
Total Fecal Weight | Days 1-9
  Total fecal weight throughout 9-day treatment period, and mean fecal weights (daily avg. of Days 5-9)
Net Balance of Potassium, Magnesium, Calcium, and Phosphorous | Days 5-9
  The net balance of cations was calculated based on dietary and fluid intake, urinary and fecal output, and emesis.
Fecal content and concentration of sodium, potassium, magnesium, calcium, phosphorous, iron, zinc, and copper | Days 5-9
Urine content and concentration of sodium, potassium, magnesium, calcium, and phosphorous | Days 5-9
Serum concentrations of sodium, potassium, magnesium, calcium, and phosphorous | Days 5-9

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Blok, MD, Principal Investigator — Jasper Clinic, Inc.
Locations (1):
- Jasper Clinic, Inc., Kalamazoo, Michigan, United States

REFERENCES:
- [Derived] Henderson LW, Dittrich HC, Strickland A, Blok TM, Newman R, Oliphant T, Albrecht D. A Phase 1 dose-ranging study examining the effects of a superabsorbent polymer (CLP) on fluid, sodium and potassium excretion in healthy subjects. BMC Pharmacol Toxicol. 2014 Jan 25;15:2. doi: 10.1186/2050-6511-15-2. PMID 24460668